CLINICAL TRIAL: NCT02771522
Title: Monitoring of Caries Lesion Activity in Orthodontic Patients With the Calcivis System
Brief Title: Caries Lesion Activity in Orthodontic Patients - Calcivis System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calcivis Ltd (Industry)
Collaborators: Medsource UK Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAL-03-2015
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-06

CONDITIONS: Dental Caries
Keywords: Caries, Acitivity, Demineralsiation
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active post-othodontic lesions (Other): Imaging with the Calcivis System
  Interventions: Device: Calcivis System

INTERVENTIONS:
Device: Calcivis System — Following de-bond, and identification of active post-orthodontic white spot lesions at baseline with the Calcivis System, each active tooth will be again be imaged at 2, 4, 8 and 12 weeks. Both black & white and luminescent images images of the teeth are taken. The images of each tooth are overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
  Other Names: Calcivis Caries Activity Imaging System

SUMMARY:
This is a prospective, single-centre clinical study to monitor caries lesion activity in orthodontic patients with the Calcivis System over a 12 week period. Dentists will identify patients who have had dental appliances in place for a minimum of 12 months and have visible white spot lesions on the anterior surfaces of incisors and / or canines at de-bond. Following de-bond, images of the tooth surface will be taken with the Calcivis System. Presence or absence of elevated luminescence on the images will indicate activity / inactivity. Only patients with at least one tooth identified as active with the Calcivis System will continue in the study and be followed up at 2, 4, 8 and 12 weeks de-bond. Images of the active teeth will be taken with the Calcivis System as before, at each follow-up visit.

The percentage of teeth showing luminescence using the Calcivis System will be calculated and summarised for all subjects for each post-baseline visit, and additionally by Investigator. This will then be summarised over all subjects for each post-baseline visit.

DETAILED DESCRIPTION:
Dental caries (tooth decay) is a significant clinical and public health problem. The development of caries lesions involves a net mineral loss of dental tissue, which can lead to progressive loss of tooth structure and associated pain and disease. Detecting, assessing, diagnosis and treating such lesions are core activities in dentistry. Currently the main detection and diagnosis aids are visual inspection and the used of a probe, together with X-ray images. Determination of the activity status of a lesion (how likely it is to progress) is requires to assess treatment needs. Currently methods are problematic and involve the clinicians' subjective assessment and / or monitoring of lesions progression over a number of visits.

It is generally recognised and reported in the dental literature that patients undergoing orthodontic treatment with fixed appliances find it difficult to maintain meticulous oral hygiene and that, as a result, plaque accumulates adjacent to the orthodontic brackets (which are usually placed on the buccal, Free Smooth, surfaces of teeth, which are readily visible) holding the metal wires which are involved in moving the teeth - thus white spot lesions commonly develop at these sites of plaque stagnation. These lesions are, de facto, actively developing during orthodontic treatment, thus represent 'active lesions'. Once the wires and brackets are removed post-treatment, normal oral hygiene can be resumed, the plaque/biofilm over these lesions is readily removed and they become arrested, i.e. the demineralisation process ceases. Thus during a short period of time - a matter of weeks - there is usually a transition from active to inactive status for these 'orthodontically-induced' white spot lesions. By assessing and monitoring these lesions, using the Calcivis device, at relatively short intervals during this period of lesion status transition immediately post orthodontic treatment it would be possible to monitor the reduction in the demineralisation process as these lesions arrest.

A previous clinical study on the prototype of the Calcivis System has been conducted. The results concluded that the Calcivis System was safe for use and the level of agreement between elevated luminescence and areas of expected activity was above 70% and not due to chance (NCT02098304).

This prospective, single-centre clinical study has been designed to assess the use of the Calcivis System for monitoring the activity levels of post-orthodontic treatment white spot lesions over time. The Dentist will share the images with the patient

The device under evaluation comprises a hand-held customized intra-oral camera which takes both black & white and luminescent images of a lesion on a tooth surface while simultaneously applying a photoprotein solution. The photo-protein detects free calcium ions on the tooth surface and produces a light signal if the caries lesion is active.

For the study, patients attending routine Orthodontic appointments to have their appliances checked, and who are identified by the Investigator as meeting the Inclusion and Exclusion criteria, and are ready for de-bond, will be approached to discuss their possible participation in the study.

Patients will be given a Patient Information Sheet to read and time to consider their participation in the study. If they are happy to participate they will asked to attend for five Study Visits - de-bond (baseline), 2, 4, 8 and 12 weeks. Written informed consent will be taken before any study procedures are conducted. As children under the age of 16 are included in this study, parent / guardian consent will be taken where appropriate.

At study Visit 1, demographics, relevant medications, oral hygiene and orthodontic history data will be collected.

The orthodontist will carry out an oral examination and the tooth / teeth identified as per inclusion / exclusion criteria, will be cleaned with prophy paste, rinsed with tap water and a 3-in-1 air / water spray before being air dried and staged as per ICDAS coding. Reference intra-oral photographs will be taken of each tooth. The free smooth tooth surfaces will again be air dried before taking the black & white and luminescent images with the Calcivis System. After imaging is completed, patients rinse out with tap water. Adverse event will be collected throughout. The dentist will then share the images of the teeth with the patient. Post imaging questionnaires will be completed by each patient at the end of Study Visit 1 and user questionnaires completed by the dental team at the end of each Study Visit 1 day.

Only patients who have 'active' lesions on de-bond, as confirmed with the Calcivis System at the baseline visit, will be followed up in this study. If all lesions are assessed as 'inactive', the patient will be withdrawn from the study

Eligible patients will return for Study Visits at 2, 4, 8 and 12 weeks post-de-bond. At each of these visits, following a reference photograph of the teeth, each tooth which was "active" at Study Visit 1 will again be imaged with the Calcivis System as described above and the images shared with the patient. In addition, both Patient and User Questionnaires will be completed at the final Study Visit at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 12 years old
2. Patient must have had orthodontic appliances placed on the upper incisors and / or canines for at least 12 months, and be ready for de-bond
3. Patient must have at least one, active white spot lesion identified by the Calcivs System immediately post de-bond
4. Patient and / or parent or guardian must be willing and able to give written informed consent
5. Patient and / or parent or guardian must be willing and able to adhere to study schedule

Exclusion Criteria:

1. Any Patient with recent tooth bleaching (within previous two weeks of imaging with the Calcivis System) or within the follow-up period
2. Any patient currently taking part in a clinical research study, or who has taken part in a clinical research study in the previous three months
3. Pregnant and / or nursing mothers

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aman Ulhaq, BDS, MFDS, MSc, MOrtho, Study Director — Edinburgh Dental Institutie; Niall McGuinness, FDS, MOrth, MSCD, DDS, PhD, Principal Investigator — Edinburgh Dental Institute; Eamon Howard-Bowles, BDS, MFDS, PG Cert, Principal Investigator — Edinbuirgh Dental Institute
Locations (1):
- Edinburgh Dental Institute, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by two Investigators from a routine NHS Orthodontic clinic between 15 February 2017 and 01 May 2018.
  Of the 36 patients attending Visit 1, 30 were eligible for Calcivis imaging ( 3 patients were pregnant, 2 patients had appliances on less than 12 months and I patient did not have visible white spot lesions).
Units Other Than Participants: Teeth
Groups:
- Active Post-othodontic Lesions: Following de-bond, and identification of active post-orthodontic white spot lesions at baseline with the Calcivis imaging system, active teeth were again imaged at 2, 4, 8 and 12 weeks.
  Black & white and luminescent images of the teeth were taken. The images of each tooth were overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Period: Overall Study
Arm/Group | Active Post-othodontic Lesions
Started (Patients attending baseline visit at de-bond and imaged with Calcivis System) | 30; 119 Teeth (119 teeth imaged with the Calcivis System from 30 patients)
Completed (Patients attending final visit at 8 weeks post de-bond and imaged with Calcivis System) | 22; 87 Teeth (87 teeth imaged with the Calcivis System fro 22 patients)
Not Completed | 8; 32 Teeth
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2
Not completed — No white spot lesions | 3

BASELINE CHARACTERISTICS:
Population: Of the 30 patients, 119 teeth were imaged
Groups:
- Active Post-othodontic Lesions: Imaging with the Calcivis System: Following de-bond, and identification of active post-orthodontic white spot lesions at baseline with the Calcivis imaging system, each active tooth was again be imaged at 2, 4, 8 and 12 weeks. In order to improve study recruitment, a Protocol Amendment was approved to reduce the overall number of visits to 2, 4 and 8 weeks, however there is data available form all time points.
  The images of the teeth are taken immediately before and after application of a small amount of solution. The images of each tooth are overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Active Post-othodontic Lesions
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — All patients who had teeth imaged
  years | 19.9 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30
Number of teeth imaged and deemed active [Number; unit: Teeth] — Number of teeth imaged by CALCIVIS imaging device deemed active
  Teeth | 73

OUTCOME MEASURES:

1. Primary Outcome: Presence or Absence of Elevated Luminescence
Description: Percentage of active teeth showing luminescence (as measured by Calcivis System imaging) over time
Time Frame: 0, 2, 4, 8 and 12 weeks
Population: From 30 participants a total of 119 teeth were imaged at baseline then different numbers of patients attended different follow-up visits
Measure: Number; unit: % active teeth with luminescence
Units Other Than Participants: Teeth
Groups:
- Active Post-othodontic Lesions: Imaging with the Calcivis System - Percentage teeth with luminescence over time
Arm/Group | Active Post-othodontic Lesions
Number analyzed (Participants) | 30
Number analyzed (Teeth) | 119
% active teeth with luminescence
  Baseline | 61.7
  2 weeks post de-bond: number analyzed (Participants) | 13
  2 weeks post de-bond: number analyzed (Teeth) | 51
  2 weeks post de-bond | 17.3
  4 weeks post de-bond: number analyzed (Participants) | 21
  4 weeks post de-bond: number analyzed (Teeth) | 83
  4 weeks post de-bond | 6.0
  8 weeks post de-bond: number analyzed (Participants) | 22
  8 weeks post de-bond: number analyzed (Teeth) | 87
  8 weeks post de-bond | 10.2
  12 weeks post de-bond: number analyzed (Participants) | 8
  12 weeks post de-bond: number analyzed (Teeth) | 31
  12 weeks post de-bond | 6.3

2. Primary Outcome: Presence or Absence of Elevated Luminescence
Description: Percentage of active teeth showing luminescence (as measured by Calcivis System imaging) over time, per Investigator
Time Frame: 0, 2, 4, 8 and 12 weeks post de-bond
Population: From a total of 30 participants (28 patients from Investigator 1, and 2 patients from Investigator 2) a total of 119 teeth were imaged at baseline then different numbers of patients attended different follow-up visits
Measure: Number; unit: % active teeth with luminescence
Units Other Than Participants: Teeth
Groups:
- Post-orthodontic Lesions: Imaging with the Calcivis System - Percentage teeth with luminescence over time, per Investigator
Arm/Group | Post-orthodontic Lesions
Number analyzed (Participants) | 30
Number analyzed (Teeth) | 119
% active teeth with luminescence
  Site 11 - Baseline: number analyzed (Participants) | 28
  Site 11 - Baseline: number analyzed (Teeth) | 112
  Site 11 - Baseline | 58.9
  Site 11 - 2 weeks post de-bond: number analyzed (Participants) | 11
  Site 11 - 2 weeks post de-bond: number analyzed (Teeth) | 44
  Site 11 - 2 weeks post de-bond | 11.4
  Site 11 - 4 weeks post de-bond: number analyzed (Participants) | 19
  Site 11 - 4 weeks post de-bond: number analyzed (Teeth) | 76
  Site 11 - 4 weeks post de-bond | 2.6
  Site 11 - 8 weeks post de-bond: number analyzed (Participants) | 20
  Site 11 - 8 weeks post de-bond: number analyzed (Teeth) | 80
  Site 11 - 8 weeks post de-bond | 6.3
  Site 11 - 12 weeks posar de-bond: number analyzed (Participants) | 6
  Site 11 - 12 weeks posar de-bond: number analyzed (Teeth) | 24
  Site 11 - 12 weeks posar de-bond | 8.3
  Site 31 - Baseline: number analyzed (Participants) | 2
  Site 31 - Baseline: number analyzed (Teeth) | 7
  Site 31 - Baseline | 100.0
  Site 31 - 2 weeks post debond: number analyzed (Participants) | 2
  Site 31 - 2 weeks post debond: number analyzed (Teeth) | 7
  Site 31 - 2 weeks post debond | 50.0
  Site 31 - 4 weeks posat de-bond: number analyzed (Participants) | 2
  Site 31 - 4 weeks posat de-bond: number analyzed (Teeth) | 7
  Site 31 - 4 weeks posat de-bond | 37.5
  Site 31 - 8 weeks post de-bond: number analyzed (Participants) | 2
  Site 31 - 8 weeks post de-bond: number analyzed (Teeth) | 7
  Site 31 - 8 weeks post de-bond | 50.0
  Site 31 - 12 weeks post de-bond: number analyzed (Participants) | 2
  Site 31 - 12 weeks post de-bond: number analyzed (Teeth) | 7
  Site 31 - 12 weeks post de-bond | 0.0

3. Secondary Outcome: Number of Non-patient Related Adverse Events With the Calcivis System
Description: All adverse events and device deficiencies were collected throughout the study on Adverse Event Forms
Time Frame: 0 days, 2, 4, 8 and 12 weeks
Population: All patients imaged with the Calcivis System
Measure: Number; unit: Non-patient-related Adverse Events
Groups:
- Active Post-othodontic Lesions: Imaging with the Calcivis System: Following de-bond, and identification of active post-orthodontic white spot lesions at baseline with the Calcivis System, each active tooth will be again be imaged at 2, 4, 8 and 12 weeks. Black & white and luminescent images of the teeth were taken. The images of each tooth are overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Active Post-othodontic Lesions
Number analyzed (Participants) | 30
Non-patient-related Adverse Events | 3

4. Secondary Outcome: Patient Experience
Description: Completion of Patient Questionnaires after imaging with the Calcivis System
Time Frame: Baseline
Population: Patient Questionnaires comprised of two questions and patients were asked to tick the most appropriate response on a three-point scale
Measure: Number; unit: participants
Groups:
- Post-orthodontic Lesions: Imaging with the Calcivis System -Following de-bond, and identification of active post-orthodontic white spot lesions at baseline with the Calcivis System, each active tooth will be again be imaged at 2, 4, 8 and 12 weeks. Black & White and luminescent images were taken. he images of each tooth are overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Post-orthodontic Lesions
Number analyzed (Participants) | 30
participants
  Calcivis System experience:good | 27
  Calcivis System experience:neither good nor bad | 3
  Calcivis System experience:bad | 0
  Calcivis System - seeing images:helpful | 30
  CalcivisSystem-images-neither good nor bad | 0
  CalcivisSystem - seeing images - bad | 0

5. Secondary Outcome: Patient Experience
Description: Completion of Patient Questionnaires after imaging with the Calcivis System at patient's final visit
Time Frame: Final Visit - either 8 or 12 weeks post debond
Population: Patient Questionnaires comprised two questions and patients asked to tick the most appropriate response on a three-point scale
Measure: Number; unit: Participants
Groups:
- Post-orthodontic Lesions: Imaging with the Calcivis System -Following de-bond, and identification of active post-orthodontic white spot lesions at baseline with the Calcivis System, each active tooth will be again be imaged at 2, 4, 8 and 12 weeks. Black & White and luminescent images were taken. The images of each tooth are overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Post-orthodontic Lesions
Number analyzed (Participants) | 18
Participants
  Calcivis System experienc: good | 16
  Calcivis System experience: neither good nor bad | 2
  Calcivis System experience: bad | 0
  Calcivis System-seeing images: helpful | 18
  CalcivisSystem images:neitherhelpfuln | 0
  Calcivis System - seeing images: unhelpful | 0

6. Secondary Outcome: User Questionnaires
Description: Completion of User Questionnaires after imaging with the Calcivis System
Time Frame: Baseline visit
Population: User Questionnaires were completed by the dentist and nurse at the end of every imaging session about their experiences using the Calcivis System. They were asked to tick the most appropriate response on a three-point scale e.g. easy, neither easy nor difficult , difficult.
Measure: Number; unit: User Questionniares
Units Other Than Participants: Questionnaires
Groups:
- Active Post-othodontic Lesions: Imaging with the Calcivis System -
  User Questionnaires comprised four questions and users were asked to tick the most appropriate response on a three-point scale
Arm/Group | Active Post-othodontic Lesions
Number analyzed (Participants) | 30
Number analyzed (Questionnaires) | 30
User Questionniares
  Calcivis System preparation:easy | 21
  CalcivisSystempreparation:neithereasynordifficult | 9
  Calcivis system preparation: difficult | 0
  Calcivis System use: easy | 17
  Calcivis System use: neither easy nor difficult | 11
  calcivis System use: difficult | 2
  Calcivis System experience: good | 24
  Calcivis System experience:neither good nor bad | 4
  Calcivis System experience: bad | 2
  Understand instructions:easy | 19
  Understand instructions:neither easy nor difficult | 11
  Understand instructions: difficult | 0

ADVERSE EVENTS:
Time Frame: 12 weeks post baseline visit
Description: All adverse events and device deficiencies were collected throughout the study on Adverse Event Forms
Groups:
- Active Post-othodontic Lesions: Imaging with the Calcivis System: Following de-bond, and identification of active post-orthodontic white spot lesions at baseline with the Calcivis System, each active tooth will be again be imaged at 2, 4, 8 and 12 weeks. The images of the teeth are taken immediately before and after application of a small amount of disclosing solution. The images of each tooth are overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Active Post-othodontic Lesions
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Post-othodontic Lesions (N=30)
non patient related adverse events (Product Issues) | 3 (3) — Term from definition in ISO14155:2011 (E) Device Deficiency - inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT02771522/SAP_000.pdf
  • Study Protocol (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT02771522/Prot_001.pdf